CLINICAL TRIAL: NCT00001368
Title: Cytokine and Leukocyte Activation Profile as a Risk Factor for Cerebral Vascular Disease and Stroke
Brief Title: Potential Risk Factors for Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930220; 93-N-0220
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-11

CONDITIONS: Carotid Atherosclerosis; Cerebrovascular Accident; Diabetes Mellitus; Hypercholesterolemia; Hypertension
Keywords: Cerebral Ischemia; Hypertension; Immune Response; Carotid Stenosis; Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases; Stroke; Diabetes Mellitus; Hypercholesterolemia; Hypertension; Brain Ischemia; Carotid Stenosis; Atherosclerosis | interventions — Cytokines

INTERVENTIONS:
Procedure: cytokine and leukocyte activation profile

SUMMARY:
Early studies have shown that the immune system may play a role in the development of strokes. Conditions such as high blood pressure, high cholesterol, diabetes, and old age can activate the immune system and increase the risk of developing hardening of the arteries (atherosclerosis) and damaged blood vessels.

Researchers will attempt to characterize factors that may contribute to atherosclerosis and stroke by measuring certain components of the immune system, cytokines and leukocyte activation. Measurements will be taken from patients that are considered to be stroke prone and from patients without risk factors for the development of stroke. Researchers will measure the immune system components at the beginning of the study, at six months, and at the one-year completion of the study.

The study will attempt to determine;

I) If patients with risk factors for stroke have an increased activation of the immune system

II) If patients with risk factors for stroke that are symptomatic have higher levels of immune system activation compared to patients who do not have symptoms

III) If patients with increased activation of the immune system have accelerated hardening of the arteries (atherosclerosis)

DETAILED DESCRIPTION:
Preliminary studies indicate that activation of the immune system by risk factors for stroke (hypertension, hypercholesterolemia, diabetes and age) increases the risk of atherosclerosis and the formation of intravascular thrombosis. By measuring the levels of cytokine and leukocyte activation in the stroke prone population and age matched controls without risk factors, an attempt will be made to characterize those factors which potentially increase the risk for carotid atherosclerosis and subsequent cerebral infarctions.

A total of one hundred twenty subjects with risk factors for stroke and forty controls will be enrolled over a two year period and followed for one year. All subjects will have blood drawn at the time of enrollment, at six months, and one year to measure cytokine levels (including Interleukin-I, Tumor Necrosis Factor-Alpha, Interleukin-8) and leukocyte activation/receptor (including Intercellular Adhesion Molecule-1 (ICAM-1), Endothelial Leukocyte Adhesion Molecule-1 (ELAM-1), V-Cell Adhesion Molecule (VCAM), and Macrophage Antigen-1). Carotid dopplers will be performed at the time of enrollment and at one year.

An analysis will be performed to: 1) determine if patients with risk factors for stroke have an increased activation of baseline cytokine levels and leukocytes, 2) determine if patients who have stroke risk factors and are symptomatic have an increased activation of cytokines and leukocyte vs. asymptomatic patients, and 3) determine if patients with increased cytokine/leukocyte activity have accelerated atherosclerosis of the carotid arteries.

ELIGIBILITY:
Male or female greater than 18 years of age.

Patient must have documented hypertension (diastolic BP greater than 90 mmHg or systolic BP greater than 140 mmHg) for greater than 1 year OR hypercholesterolemia (LDL greater than 160 or total Chol greater than 240 with a total cholesterol/HDL-Chol ratio more than 1.6 for greater that 1 year OR Diabetes (blood glucose greater than 150 mg/dl requiring oral antihyperglycemics or insulin dependent) for greater than 1 year OR any combination.

Subgroup eligibility for risk factors with cerebral ischemic events must meet criteria #2 plus documented stroke by physical exam and CT and/or MRI consistent with ischemic infarction or TIA witnessed and recorded by medical personnel.

Patient will be excluded if enrollment time is within 30 days of a stroke, myocardial infarction, or surgery. Patient may be enrolled after 30 days of the above events.

No patients on immunosuppressive therapy.

No patients who are unable to follow up for 1 year from the time of enrollment.

No stroke patients with an identifiable cardiac source (including atrial fibrillation, mural thrombus, valvular disease with vegetation).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 1993-10; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] DeGraba TJ. The role of inflammation after acute stroke: utility of pursuing anti-adhesion molecule therapy. Neurology. 1998 Sep;51(3 Suppl 3):S62-8. doi: 10.1212/wnl.51.3_suppl_3.s62. PMID 9744839
- [Background] Siren AL, Heldman E, Doron D, Lysko PG, Yue TL, Liu Y, Feuerstein G, Hallenbeck JM. Release of proinflammatory and prothrombotic mediators in the brain and peripheral circulation in spontaneously hypertensive and normotensive Wistar-Kyoto rats. Stroke. 1992 Nov;23(11):1643-50; discussion 1650-1. doi: 10.1161/01.str.23.11.1643. PMID 1440713
- [Background] Loddick SA, Wong ML, Bongiorno PB, Gold PW, Licinio J, Rothwell NJ. Endogenous interleukin-1 receptor antagonist is neuroprotective. Biochem Biophys Res Commun. 1997 May 8;234(1):211-5. doi: 10.1006/bbrc.1997.6436. PMID 9168991